CLINICAL TRIAL: NCT00596531
Title: Clinical Trial of Acamprosate for Tinnitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, William Hal Martin, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00003412; IRB00003412
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Tinnitus
Keywords: Tinnitus; acamprosate; clinical trial
MeSH Terms: conditions — Tinnitus | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Subjects will take acamprosate (Campral) at a dose of 666 mg. three times daily (morning, lunch time, bed time) for 28 days. Only responders will be included in the subsequent double-blind cross over arms after a minimum washout period of 4 weeks.
  Subjects will randomly be assigned to Group 1 (A/B) or Group 2 (B/A) after completion of Phase I and its subsequent washout period (Figure 1, periods 1 and 2). Group 1 will receive acamprosate (Campral) at a dose of 666 mg. three times daily for 24 weeks followed by a 4-week washout period
  Interventions: Drug: Acamprosate
- B (Placebo Comparator): Group 2 will be assigned to the placebo group and take matched placebos for next 24 weeks followed by a 4-week washout period. After the washout period each group will be assigned to the other intervention (acamprosate or placebo) and complete another trial for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acamprosate — Oral administration, 666 mg, tid, for 4 months
  Other Names: Campral
  Arms: A
Drug: Placebo — Oral administration of 2 pills, tid, for 4 months
  Arms: B

SUMMARY:
The objective of this project is to determine whether acamprosate is more effective at providing relief for tinnitus than a placebo.

Acamprosate has been suggested to be effective in reducing tinnitus annoyance in a preliminary study. Study evidence indicates that tinnitus is related to increased excitatory spontaneous brain activities. Acamprosate may help restore the excitatory/inhibitory balance in the brain and thus reduce tinnitus.

The current study includes three phases. The first phase is an open-label screening study used to identify tinnitus subjects responding to acamprosate. These responding subjects will enter the second phase, which is a double blind, placebo-controlled study aimed at confirming the subjects' responses to acamprosate. In the third phase, clinical parameters of both responders and non-responders will be compared using a multi-linear regression model to determine characteristics that define the sub-group of tinnitus patients that are likely to benefit from acamprosate treatment. Participation in the study requires that individuals come to Portland, Oregon at least 6 times over 16 months for evaluation and data collection.

DETAILED DESCRIPTION:
The current study includes three phases. The first phase is an open-label screening study used to identify tinnitus subjects responding to acamprosate. These responding subjects will enter the second phase, which is a double blind, placebo-controlled study aimed at confirming the subjects' responses to acamprosate. In the third phase, clinical parameters of both responders and non-responders will be compared using a multi-linear regression model to determine characteristics that define the sub-group of tinnitus patients that are likely to benefit from acamprosate treatment. Participation in the study requires that individuals come to Portland, Oregon at least 6 times over 16 months for evaluation and data collection.

Measurements: Subjects will be brought in for baseline evaluation for Phase II four weeks after finishing their course of acamprosate during Phase I. Subjects will receive a full audiometric evaluation. Subjects with active otologic disease at that time will be excused. Tinnitus pitch and loudness matching per Johnson and Goodwin, (1981) will be performed noting octave confusion. Loudness matching will be performed using a 1 kHz tone presented to the ear contralateral to the tinnitus of interest to minimize complications tinnitus was often too high a level to test (beyond the limits of the equipment). This problem occurs less often when using a 1 kHz comparison tone because most subjects have reasonable auditory thresholds at that frequency. Minimum masking levels (MML) will be determined by measuring the level at which a 2 kHz to 12 kHz band of noise completely masks the tinnitus in the ipsilateral ear. Residual inhibition or post-masking change testing will be conducted at the end of the tinnitus testing. The 2 kHz to 12 kHz band of noise will be elevated to 10 dB above the MML (if tolerable) and remain on continuously in the ear ipsilateral to the tinnitus for 60 seconds. At that point, the masking will be turned off and the subject will be asked to identify any changes in their perceived tinnitus. If partial or complete residual inhibition occurs, their duration will be timed with a stopwatch and recorded. Subjects will also be instructed to complete VAS scores for tinnitus loudness and annoyance, the Tinnitus Handicap Inventory (THI; Newman et al, 1996) which is a 25-item questionnaire that is currently the most widely used estimator of the impact of tinnitus on an individual daily life, and the Maudsley Obsessional-Compulsive Inventory (MOCI; Rachman and Hodgson, 1980) questionnaire, which will not be used as a primary outcome measurement, but will be used in the multiple linear regression analysis of Phase III. Upon completing Phase II of the study, the subjects who do not experience improvements in their tinnitus from acamprosate will be given information about other tinnitus management options and given the opportunity to be evaluated and managed at the OHSU Tinnitus Clinic.

The primary outcome measures for Phase II will include:

Rated tinnitus loudness: VAS scores for tinnitus loudness Rated tinnitus loudness: VAS scores for tinnitus annoyance Tinnitus Severity: Tinnitus Handicap Index Matched tinnitus loudness: Loudness match re: 1kHz tone in the contralateral ear to tinnitus (unless subject has bilateral or unilateral profound hearing loss) Minimum Masking Level: MML with broad band noise in ipsilateral ear to tinnitus (unless subject has bilateral or unilateral profound hearing loss) The Prototype 2 of the Tinnitus Functional Index is a 30-question evaluation tool currently under development with funding from the Tinnitus Research Consortium through a multi-center study hosted by the OHRC. The TFI will serve as a secondary outcome measure of tinnitus severity in Phases II and III. Thus far in development, the TFI has demonstrated good reliability, validity and high sensitivity to measuring treatment-related changes in tinnitus severity (responsiveness). The TFI has not been published, but the investigators believe that it would be beneficial to this study and provide an opportunity to use the TFI in a new clinical setting.

The primary outcomes measures and the MOCI and TFI will be recorded five times during the study: At the baseline visit (Figure 1, beginning of period 3), at the end of the first 24 weeks (between periods 3 and 4), at the end of the wash out period (between periods 4 and 5), at the end of the second 24-week period (end of period 5) and 4 weeks after the completion of the Phase I trial. All audiometric and tinnitus measures and the questionnaire scores will be entered into the PATS data base.

Short-term vs. long-term measures: Tinnitus loudness matching and MML measures provide quantitative measures about the immediate status of a subject's tinnitus. Loudness and annoyance are more integrative, depending on the subject's perception of the tinnitus, but are still reflective of the immediate tinnitus conditions of the subject. THI and TFI quantify the direct and indirect impact of the tinnitus on the individual. These tools evaluate tinnitus effects that are often cumulative over long periods of time (e.g. depression, insomnia, changes in social interactions). Medications that alter brain chemistry may have an impact on either or both short and long-term tinnitus measures so both categories are being evaluated.

Treatment: Subjects will randomly be assigned to Group 1 (A/B) or Group 2 (B/A) after completion of Phase I and its subsequent washout period (Figure 1, periods 1 and 2). Group 1 will receive acamprosate (Campral) at a dose of 666 mg. three times daily for 24 weeks followed by a 4-week washout period and then by taking matched placebos for next 24 weeks. Group 2 will receive placebo for 24 weeks followed by a washout and 24 week acamprosate trial. The experiment will be double-blinded. The subjects will know that they could be taking either a placebo or acamprosate. To insure subjects are blind to the intervention, the Campral will be placed in identical capsules to those used for the cellulose placebos that will be produced for the study.

Data acquisition: VAS sheets will be completed during the initial Phase II baseline visit and 6 sets of time/dated sheets (one for loudness, one for annoyance, plus two spare sheets) will be sent home with subjects. Equivalent sets of the THI, TFI and MOCI will be included with the VAS sheets and subjects given instruction (verbally and in writing) on how to complete and return all data sheets in self-addressed stamped envelopes. Sheet acquisition will follow the course that it did in Phase I, however, they will only be collected monthly instead of weekly. The subject will return to the clinic after 24 weeks for testing including VAS, THI, TFI and MOCI evaluations. At that time they will receive their supply of capsules (medication or placebo) and new sets of VAS, THI and MOCI sheets and mailing envelopes for the second period of Phase II (Figure 1, period 5).

Psychoacoustic measures of tinnitus will be measured during the baseline visit, during the 24-week return visit, and at the conclusion of the 52-week study.

ELIGIBILITY:
Inclusion Criteria:

* Concurrent treatments: Amplification, sound generators or cochlear implants are permitted, provided they have been in use for at least one year. A four-week washout from any other tinnitus treatment or management program is required prior to entering this study.
* Hearing function: All levels of hearing function can be included recognizing that profound, bilateral losses will not be able to perform psychophysical tinnitus and hearing tests but will be able to rate subjective loudness, annoyance and impact on life.
* Tinnitus etiology: All forms of tinnitus etiology will be accepted into Phase I providing they meet the following tinnitus criterion. Duration: 1 year or longer. Stability: Constant. Severity: > 50th percentile of OHSU Tinnitus Patients based upon Tinnitus Functional Index scores. Rated loudness: >6 on a 0-10 visual numerical scale. Tinnitus location: Unrestricted.

Exclusion Criteria:

* Medical conditions: Active neurologic or otologic disease processes that may impact tinnitus perception. Auto-immune diseases. Pregnancy or planned pregnancy during the study.
* Renal function: Subjects with documented renal disorders will be excluded if renal function has creatinine clearance is <50 mL/minute.
* Digestive tract problems: Subjects with digestive tract disorders will be excluded.
* Psychological status: Beck Depression Inventory score of greater than 15.
* Tinnitus duration: Less than 1 year. Stability: pulsatile, intermittent, varying to a high degree in loudness or changing in location of perception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Index Tinnitus Functional Index Tinnitus loudness score on visual numerical scale | 15 months

SECONDARY OUTCOMES:
Depression Inventory Psychoacoustic measures of tinnitus | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: William H Martin, Ph.D., Principal Investigator — Oregon Health and Science University; Yongbing Shi, M.D., Ph.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

REFERENCES:
- See also: website for host of study — http://www.ohsu.edu/ohrc/tinnitusclinic